CLINICAL TRIAL: NCT00877318
Title: Cardiac Rehabilitation of Heart Failure Patients by Telemedicine: a Randomized Multicenter Study.
Brief Title: Cardiac Rehabilitation of Heart Failure Patients by Telemedicine
Acronym: READ
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: insufficient recruitment
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B80908-20
Record Dates: First submitted 2009-04-06; First posted 2009-04-07 (Estimated); Last update posted 2016-03-18 (Estimated); Status verified 2016-03

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Program of cardiac rehabilitation introduced in complete hospitalization pursued in day hospital during 3 months
- telemedicine (Experimental): Program of cardiac rehabilitation introduced in complete hospitalization pursued at home via a terminal during 3 months
  Interventions: Device: SCAD information system

INTERVENTIONS:
Device: SCAD information system — Cardiac rehabilitation at home by telemedicine
  Arms: telemedicine

SUMMARY:
The purpose of the READ study is to compare the continuation of the cardiac rehabilitation at home with clinical follow-up, therapeutic education, and advice on the training at the stamina, via telemedicine with the classic strategy in day hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a dysfunction of left ventricle with ejection fraction of left ventricle < 40 % appreciated by echocardiogram at hospital discharge for cardiac rehabilitation.

Exclusion Criteria:

* Patient non authorized to follow an effort training
* Therapeutic education impossible
* Pregnant woman or breast-feeding
* No assent
* Incapacity to use the terminal
* Minor patient or under supervision

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2009-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Variation of VO2 peak at 3 months in comparison to VO2 peak at hospital discharge | 3 months

SECONDARY OUTCOMES:
VO2 peak at 3 months compared with VO2 peak at the beginning of the hospitalization | 3 months
BNP | 3 months
% patient with a BNP < 300 pg/ml | 3 months
Medical treatment by ACE inhibitor (in % of target dose) | 3 months
Ejection fraction of left ventricle | 3 months
Disease knowledge questionnaire | 3 months
Life quality questionnaire (Minnesota) | 3 months
Beck questionnaire | 3 months
Day number at hospital | 3 months
Number of medical consultation | 3 months
Pharmaco-economic analysis | 3 months
Total mortality | 3 months
Cardiovascular mortality | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Annette Belin, MD, Principal Investigator — University Hospital, Caen; Rémi Sabatier, MD, Principal Investigator — University Hospital, Caen
Locations (2):
- France (2):
  - Centre Hospitalier de la Côte Fleurie, Cricquebœuf
  - William Harvey Center, Saint-Martin-d'Aubigny